CLINICAL TRIAL: NCT03641625
Title: Effect of Muscular Tissue Oxygen Saturation-Guided Management During Laparoscopic Hysterectomy on Postoperative Nausea and Vomiting: A Randomized Controlled Trial (iMODIPONV)
Brief Title: Effect of SmtO2 Guided Care on PONV (iMODIPONV)
Acronym: iMODIPONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: The Second Hospital of Hebei Medical University (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); Shandong Provincial Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); Beijing Obstetrics and Gynecology Hospital (Other)
Responsible Party: Principal Investigator, Lingzhong Meng, Professor and Division Chief, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RCT_SmtO2_PONV
Record Dates: First submitted 2018-07-27; First posted 2018-08-22 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Nausea and Vomiting; Hysterectomy; Tissue Oxygenation; Cardiac Output Management; Blood Pressure Management
Keywords: Postoperative Nausea and Vomiting; Laparoscopic Hysterectomy; Muscular Tissue Oxygen Saturation; Hemodynamic Management
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: International, multi-center, pragmatic, randomized controlled (1:1 ratio) trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Both patients and outcomes assessor are blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): In addition to usual care during surgery, the intraoperative management will be additionally managed based on the guidance of muscular tissue oxygen saturation and non-invasive hemodynamic monitoring.
  Interventions: Device: Muscular tissue oxygen saturation guided care
- Control (No Intervention): Patients will receive the usual care. Muscular tissue oxygen saturation and non-invasive hemodynamic monitoring will be used but blinded to care givers.

INTERVENTIONS:
Device: Muscular tissue oxygen saturation guided care — Muscular tissue oxygen saturation monitored at flank and arm will be maintained > 70% (absolute measurement) and > baseline throughout the entire procedure.
  Arms: Intervention

SUMMARY:
This randomized controlled trial is to investigate if SmtO2-guided management on top of the usual care, compared with the usual care only, during laparoscopic hysterectomy significantly reduces the incidence of PONV.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) remains prevalent despite the institution of various prophylactic measures. The incidence of PONV in female patients undergoing laparoscopic gynecological surgery is up to 50% with and 70% without the administration of antiemetics, respectively. The consequences of PONV range from patient discomforts, postoperative complications, prolonged hospitalization, to increased health care costs. Among the multiple risk factors, suboptimal gastrointestinal (GI) perfusion or oxygenation may be responsible for some cases of PONV; however, this speculation remains to be confirmed.5 Optimal tissue oxygenation, the balance between tissue oxygen consumption and supply, is essential for the integrity of any tissue bed that is metabolically active. However, GI oxygenation cannot be directly and continuously monitored in patients at this time. Whether there is an organ which can be used as a surrogate of the GI system, meaning that the tissue oxygenation of this surrogate organ not only can be monitored and that it also correlates with that of the GI system, is an intriguing question. Currently, tissue oxygenation can be measured using near-infrared spectroscopy (NIRS) in patients. The recent advancements of this technology enable the accurate monitoring of the oxygenation within many tissue beds depending on the location of the oximetry probe.

The recent cohort study demonstrated that there is a close relationship between muscular tissue oxygen saturation (SmtO2) and PONV in patients undergoing robotic laparoscopic hysterectomy (manuscript accepted and in production). Multiple thresholds based on threshold, AUC, and multivariable analyses are able to differentiate the risk of PONV. The following SmtO2 thresholds were found to correlate with a reduced risk of PONV: 20% above baseline; while the following thresholds correlate with an increased risk of PONV: 5% below baseline, 15% below baseline, and 20% below baseline, < 70%, < 65%, and < 60%. Taken together, our study suggests the potential therapeutic targets for PONV prophylaxis may be to maintain SmtO2 > 70% and above baseline.

In this study, the investigators aim to investigate if intraoperative care guided by SmtO2 monitoring reduces the incidence of PONV after laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. Non-smoker
3. ASA I-III
4. Elective laparoscopic procedure involving hysterectomy

Exclusion Criteria:

1. Refuse to participate
2. Emergent surgery
3. Bowel resection planned
4. Vaginal or abdominal (open) hysterectomy
5. Chemotherapy or radiotherapy before surgery
6. Significant neuro, cognitive, or psychologic disease: stroke with neurologic deficit, dementia, schizophrenia, or any condition that makes meaningful postoperative follow-ups impossible
7. Significant cardiovascular disease: low-output cardiac failure defined as a preoperative left ventricular ejection fraction < 30%, active coronary artery disease, symptomatic valvular disease, symptomatic arrhythmia with or without pacemaker and/or AICD placement
8. Significant pulmonary disease: COPD requiring home oxygen therapy, severe asthma requiring steroid treatment, other pulmonary conditions requiring home oxygen therapy
9. Severe hepatic dysfunction being evaluated for liver transplantation or with a Child-Pugh Class C classification
10. Severe renal dysfunction requiring renal replacement therapy
11. Muscular pathologies such as dystrophy, atrophy, and weakness
12. Skin conditions incompatible with the adhesive oximetry probe (e.g., delicate or tattooed skin)
13. Current or previous smoker
14. ASA Physical Score ≥ IV

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — It is female patients whom are receiving hysterectomy.
Enrollment: 800 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV within 24 hours after surgery | up to 24 hours
  Nausea: Nausea is defined as a subjective unpleasant sensation associated with the urge to vomit.
  Retching: Retching is defined as the labored, spastic, and rhythmic contraction of chest and abdominal muscles without expulsion of gastric contents.
  Vomiting: Vomiting is defined as the forceful expulsion of any gastric contents from the mouth.
  PONV: PONV refers to the occurrence of nausea, retching, and/or vomiting.

SECONDARY OUTCOMES:
Incidence of early PONV | up to 6 hours
  The incidence of PONV during postoperative 0-6 hours. The diagnostic criteria for early PONV are the same as above (outcome 1).
Severity of postoperative pain | up to 24 hours
  Postoperative pain intensity at rest and with movement expressed using NRS 0-10 (0 = no pain; 10 = worst pain) at 2, 6, and 24 h depending on the time to discharge
Time of GI recovery | up to 48 hours
  Time to GI recovery (time to first flatus, bowel motion, and/or time to tolerate oral diet, in hours)
Overall quality of recovery based on QoR-15 questionnaire | up to 24 hours
  Postoperative quality of recovery
  (using the QoR-15 questionnaire)
  QoR-15 Questions PART A How have you been feeling in the last 24 hours? (0 to 10, where 0 = none of the time [poor] and 10 = all of the time [excellent] Q.1 Able to breathe easily Q.2 Been able to enjoy food Q.3 Feeling rested Q.4 Have had a good sleep Q.5 Able to look after personal toilet and hygiene unaided Q.6 Able to communicate with family or friends Q.7 Getting support from hospital doctors and nurses Q.8 Able to return to work or usual home activities Q.9 Feeling comfortable and in control Q.10 Having a feeling of general well-being PART B Have you had any of the following in the last 24 hours? (10 to 0, where 10 = none of the time [excellent] and 0 = all of the time [poor]) Q.11 Moderate pain Q.12 Severe pain Q.13 Nausea or vomiting Q.14 Feeling worried or anxious Q.15 Feeling sad or depressed
Time to mobilization | up to 48 hours
  Time to mobilization (time to first out-of-bed mobilization, in hours)
Score of sleep quality | up to 48 hours
  Postoperative sleep quality (using NRS 0-10 (0 = no concern at all; 10 = worst ever) for the first night or the second night if the case is finished after 6pm)
In-hospital GI complications | up to 30 days
  In-hospital GI-related composite complication (composite of ileus, obstruction, perforation, and bleeding)
Non-GI-related composite complications | up to 30 days
  Both in-hospital and 30-day non-GI-related composite complications (Complication was defined as any deviation from the normal postoperative course or organ dysfunction.[23-25] Organ-specific complications include myocardial infarction, congestive heart failure, cardiac arrest, atrial fibrillation or other types of arrhythmia, pulmonary embolus, pneumonia treated with antibiotics, respiratory failure requiring intubation, respiratory insufficiency requiring physiotherapy or oxygen therapy, stroke, transient ischemic attack, postoperative delirium or cognitive decline, renal insufficiency requiring dialysis, acute kidney injury, urinary tract infection requiring antibiotics, hepatic insufficiency, gut hypoperfusion, ileus, disseminated intravascular coagulation, and sepsis. Surgery-related complications refer to surgical site bleeding, infection, anastomotic leakage, stenosis, ischemia, or tissue necrosis.)
Length of hospital stay | up to 30 days
  Length of hospital stay, in days
Rate of ICU admission | Up to 30 days
  The percentage of patients admitted to ICU after surgery
30-day mortality | 30 days
  30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Lingzhong Meng, MD, Principal Investigator — Yale University
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data are available to the editorial office of the journal to which the manuscript is submitted upon request.

REFERENCES:
- [Background] Geng ZY, Liu YF, Wang SS, Wang DX. Intra-operative dexmedetomidine reduces early postoperative nausea but not vomiting in adult patients after gynaecological laparoscopic surgery: A randomised controlled trial. Eur J Anaesthesiol. 2016 Oct;33(10):761-6. doi: 10.1097/EJA.0000000000000491. PMID 27307217
- [Background] Gan TJ, Mythen MG. Does peroperative gut-mucosa hypoperfusion cause postoperative nausea and vomiting? Lancet. 1995 Apr 29;345(8957):1123-4. doi: 10.1016/s0140-6736(95)90857-9. No abstract available. PMID 7715373
- [Background] Meng L, Xiao J, Gudelunas K, Yu Z, Zhong Z, Hu X. Association of intraoperative cerebral and muscular tissue oxygen saturation with postoperative complications and length of hospital stay after major spine surgery: an observational study. Br J Anaesth. 2017 Apr 1;118(4):551-562. doi: 10.1093/bja/aex008. PMID 28403400
- [Derived] Zhao X, Liao K, Wang W, Xu J, Meng L. Can a deep learning model based on intraoperative time-series monitoring data predict post-hysterectomy quality of recovery? Perioper Med (Lond). 2021 Apr 6;10(1):8. doi: 10.1186/s13741-021-00178-4. PMID 33820562